CLINICAL TRIAL: NCT02550379
Title: Emotion Recognition Training for Socially Anxious Adolescents: A Randomized Controlled Trial
Brief Title: Emotion Recognition Training for Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: University of Bristol (Other)
Responsible Party: Principal Investigator, Dr. Amanda Fitzgerald, Lecturer, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-15-41-Fitzgerald
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Anxiety; Depression
Keywords: Social Anxiety; Social Phobia; Depression; Emotion Recognition Training
MeSH Terms: conditions — Anxiety Disorders; Depression; Phobia, Social | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo protocol consists of 3 phases, baseline, training, and test. The baseline phase consists of 45 trials which calculates the balance point at which the participant rates a face as 'happy' rather than 'disgusted' over a continuum of 15 faces ranging from happy through ambiguous to disgust. 3 training blocks are then administered with 30 trials per block. Behavioural feedback is given during training (correct/incorrect) based on the participant's balance point at baseline. A test phase is then administered which is identical to the baseline phase to reassess the participant's balance point. The task takes approximately 15 minutes to complete all 3 phases.
  Interventions: Other: Placebo
- Intervention (Experimental): The ER training protocol consists of 3 phases, baseline, training, and test. The baseline phase consists of 45 trials which calculates the balance point at which the participant rates a face as 'happy' rather than 'disgusted' over a continuum of 15 faces ranging from happy through ambiguous to disgust. 3 training blocks are then administered with 30 trials per block. Behavioural feedback is given during training (correct/incorrect) based on the participant's balance point however this balance point is adjusted by 2 points on the 15 face continuum to train the participant to rate more faces as 'happy'. A test phase, identical to the baseline phase, is then administered to reassess the participant's balance point. The task takes approximately 15 minutes to complete all 3 phases.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Emotion Recognition Training
  Arms: Intervention
Other: Placebo — Placebo Training
  Arms: Placebo

SUMMARY:
While it has been hypothesised that individuals who experience social anxiety are more likely to misread facial emotions as threatening or disapproving, researchers have proposed that the difficulty may lie in decoding ambiguous facial expressions rather than identifying emotions which are expressed with greater intensity. Emotion recognition (ER) training provides a promising new avenue of research which may be beneficial in altering emotion processing biases which maintain or increase symptoms of mental health disorders. This study will examine the effectiveness of ER training in a community-based sample of young people (15-18 years) who report high levels of social anxiety. The intervention aims to alter emotion processing biases through a training procedure designed to promote the perception of happiness over disgust in ambiguous facial expressions which we hypothesise will subsequently reduce symptoms of social anxiety.

The study design consists of two phases. During Phase 1 participants will complete a screening questionnaire. This questionnaire will include a measure of the affective, cognitive, and behavioural components of social anxiety in adolescence. Depending on their suitability (i.e. scoring above a cut-off on a standardised measure of social anxiety in Phase 1 of the study), participants may then be invited to take part in a 4-day computer-based emotion recognition training programme (Phase 2). The purpose of this phase is to see if ER training will help young people feel less worried or nervous in social situations by training them to interpret ambiguous facial expressions as expressing a positive emotion (happy rather than disgusted).

Participants will be randomly assigned to either the intervention or placebo (inactive) group. Both groups will be asked to complete a 4-day programme involving one computer training session per day (each session takes approximately 20 minutes). Questionnaires will also be given to participants to complete before and after the intervention, along with a 2-week follow-up assessment. These will include questionnaires to measure social anxiety, depressive symptoms, and fear of negative evaluation. Each questionnaire will take approximately 15 minutes to complete. Participants will not know whether they have received the intervention or placebo training until after the intervention.

DETAILED DESCRIPTION:
Social anxiety disorder (SAD) is among the most prevalent mental disorders in adolescence, 10% of females and 5% of males are diagnosed with SAD in adolescence. SAD is characterised by marked fear or anxiety about social situations in which the individual is exposed to possible scrutiny by others. SAD is associated with social isolation, poor social skills, low self-esteem, and future comorbid mental disorders. Social anxiety typically develops during adolescence, thus there is a need to detect and treat it early prior to the development of a clinically-diagnosed SAD. Most early interventions for social anxiety have used Cognitive Behavioural Therapy (CBT), which focuses on modifying explicit verbal cognitions. However, many adolescents do not have access to CBT and many finding it demanding.

Research suggests that individuals who have high levels of social anxiety are more likely to misread facial emotions as threatening or disapproving, and researchers have proposed that the difficulty may lie in decoding low intensity facial expressions rather than identifying facial emotions which are expressed with greater intensity. In social anxiety, a bias towards perceiving ambiguous facial expressions as negative may give rise to avoidant behaviour and maintain or increase symptoms; therefore, this emotion processing bias may be a powerful bias for researchers to target with the aim of developing interventions to reduce symptoms.

ER training provides a promising new line of research which may be beneficial in altering emotion processing biases which maintain or increase symptoms of mental health disorders. Research has shown that ER training may be effective in reducing depressive symptoms in analogue populations with high levels of depression and anger and aggressive behaviour in healthy adults and adolescent youth at high risk of criminal offending and delinquency.

Present Study:

This research tests the effectiveness of ER training in reducing social anxiety in adolescents. Given that the age of onset of social anxiety is adolescence, peaking in late teens, this research focuses on 15-18 year olds.

Aims & Objectives:

To test the effectiveness of ER training in reducing social anxiety in adolescents. The intervention aims to alter emotion processing biases through a training procedure designed to promote the perception of happiness over disgust in ambiguous facial expressions which we hypothesise will subsequently reduce symptoms of social anxiety.

Central Research Questions:

Is ER training associated with:

I. An increase in the perception of positive (happy) over negative (disgust) emotions in faces displaying ambiguous emotional expressions? II. A decrease in negative evaluations? III. A decrease in social anxiety? IV. A decrease in other forms of anxiety and/or symptoms of depression?

PHASE 1: SCREENING FOR SOCIAL ANXIETY IN ADOLESCENTS Objective: To screen for sub-clinical levels of social anxiety in adolescents. School Sampling: Approximately 8 large second-level schools in Dublin will be randomly selected from the Department of Education and Skills 2012 published list of schools.

Power Analysis: Using G*Power 3.1, the sample size was determined as 111 based on the following parameters: a medium effect size of 0.3, alpha of 0.05, power of 0.8, a repeated measures within-between interaction: 2 (Randomization) X 3 (Pre, Post, Follow-up).

Participants: Adolescents aged 15-18 years in second-level schools will be invited for the initial screening.

Procedure: Adolescents must return parental and informed consent forms. Participants will be screened using the Social Phobia and Anxiety Inventory for Children (SPAI-C). Participants scoring above the cut-off of ≥18 will be invited to participate in the intervention (Phase 2).

Approximately 440 second-level students across 8 schools will be invited to complete screening. With an approximate response rate of 50% (N=220), and using a cut-off of ≥18 120 will be identified (60 per condition).

PHASE 2: RANDOMIZED CONTROL TRIAL Objective: To compare the effectiveness of ER to placebo training in reducing social anxiety.

Participants: Adolescents from Phase 1 screening above a cut-off of ≥18 will be invited to participate in the intervention and will be randomly assigned to ER/placebo training. On the basis of screening, the PI will ensure group equivalence across ER versus placebo groups on key variables (e.g., age, gender, social anxiety) in advance of randomization. Post randomization, independent variables will be checked to ensure they are balanced across groups so as not to contaminate outcomes of the study.

Procedure:

Participants in both ER and placebo training groups will receive 4 training sessions over 4 consecutive days. The intervention will be performed on a laptop during school and delivered in a quiet room with the researcher present. Pre-intervention data will be collected on day 1 prior to training, post-intervention data will be collected on day 4 following training, with a follow-up assessment at 2-weeks post-intervention.

Training Task:

Participants will complete training over 4 consecutive days in schools. Each session will include a computerised training programme comprised of three phases, baseline, training, and test,which will take approximately 15 minutes to complete. A follow-up assessment will be completed two weeks post-intervention. During the 2-week follow-up assessment participants will complete a final assessment of emotion sensitivity using the test phase of the emotion recognition task.

* Prototypical 'happy' and 'disgust' composite images generated from 40 individual faces (20 x male, 20 x female) showing a disgust facial expression, and the same 40 individuals showing a happy expression.
* Prototypical images used as endpoints to generate a linear morph sequence that consists of images that change incrementally from unambiguously 'happy' to unambiguous 'disgust', with emotionally ambiguous images in the middle. The proposed research will include a sequence with 15 equally spaced images for each gender (male and female) for use as experimental stimuli.
* Previous research by the University of Bristol has used stimuli portraying male faces only. The task stimuli for the current research will be matched to the participant's gender, i.e. female participants will complete a task which will include female face stimuli and male participants will complete a task which will include male face stimuli.
* Baseline and test phases will consist of 45 trials, in which each of the stimuli from the morph sequence will be presented to the participant three times. The task will require the participant to make a forced choice judgement as to whether each face is displaying a happy or disgust expression. Images will be presented one at a time, in random order, for 150 milliseconds. Stimuli will be preceded by a fixation cross, which will be presented for a random period ranging from 1500 to 2500 milliseconds. Subsequent to presentation, and to prevent processing of after images, a backward mask of noise will be presented for 250 milliseconds, followed by a prompt asking the participant to respond. This will remain on screen until the participant makes response (i.e., a judgement of 'happy' or 'disgust').
* Trials in the training phase will be similar to trials in the baseline and test phases with respect to inter-trial interval and stimuli presentation, but with the addition of feedback subsequent to the participant's response. In the placebo condition, feedback will be based on the participant's baseline balance point. That is, responses will be classified as 'correct' if the participant identified images below the original balance point image as 'disgust' and above it as 'happy', and otherwise are classified as 'incorrect'. Feedback will be a message saying 'Correct / Incorrect! That face was disgust/happy'. In the training condition, feedback will be again based on the participant's baseline balance point, but the 'correct' classification will be shifted two morph steps towards the 'disgust' end of the continuum, so that the two images nearest the balance point that the participant would previously have classified as 'disgust' at baseline will be considered 'happy' when providing feedback. In each training block, each face from the 15 face continuum will be presented twice. The order of presentation will be randomized within each block. Three training blocks will be given to each participant, resulting in 90 training trials per session and a total of 360 training trials in total.

Outcome Measures:

Outcome measure will be administered to all participants in the RCT pre-intervention (baseline on day 1), post-intervention (day 4), and at 2-week follow-up, including:

Emotion Sensitivity Measurement Accuracy assessed using baseline and test measurements at each ER/placebo training session.

Social Phobia and Anxiety Inventory for Children (SPAI-C) The SPAI-C is a 26-item self-report instrument and has good psychometric properties with adolescent samples. The SPAI-C measures the somatic, cognitive, and behavioural aspects of social phobia in children and adolescents. Questions relate to how nervous the respondent feels when carrying out certain tasks and responses are rated on a 3-point scale from never, or hardly ever to most of the time, or always with higher scores indicating greater levels of social anxiety.

Brief Fear of Negative Evaluations Scale - Revised (BFNE-R) Negative evaluations are an important aspect of social anxiety. The BFNE-R is a 12-item measure which assesses fear of negative evaluation. Items are responded to on a 5-point Likert scale from 0 to 4. The BFNE-R has shown high internal consistency and correlates well with the original BFNE.

Screen for Child Anxiety Related Disorders (SCARED) Child Version The SCARED is used to screen for signs of anxiety disorders. The 41-item measure is used to measure anxiety, including panic, separation anxiety, generalised anxiety, social avoidance, and school phobia. It has shown high reliability with adolescents. Items are rated on a 3-point Likert scale. Internal consistencies have been shown to be high with adolescent samples.

Depression Subscale of the Revised Child Anxiety and Depression Scale (RCADS) The RCADS is a 47-item self-report measure and has good psychometric properties with adolescent samples. The Depression Subscale contains 10 items. Items relating to the frequency with which depressive symptoms are experienced are rated on a 4-point Likert scale.

Research Design: A mixed model 2 (Randomization) x 3 (Time) complex design combining between subjects and within subjects conditions will be employed. Each participant will be tested at pre-intervention, post-intervention, and 2-week follow-up.

Independent Variables:

Randomization (K=2; ER training/ Placebo) Time (K=3; Pre-intervention[day 1], Post-intervention [day 4], and Follow-up)

Analyses:

All analyses on change in social anxiety, anxiety, depression, and fear of negative evaluation will be conducted as intention-to-treat analyses.

Descriptive statistics Chi-square analyses and ANOVAs Primary analyses will consist of two-way repeated ANOVAs 2 (Randomization) x 3 (Time) to test the variables under study.

ELIGIBILITY:
Inclusion Criteria:

• Those who score above the cut-off on the SPAI-C

Exclusion Criteria:

* Those with a diagnosed mental health disorder
* Those who are currently attending a mental health professional
* Those scoring below the cut-off on the SPAI-C
* Those who decline to participate
* Those whose parents/guardians do not provide written consent

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in social anxiety at post-intervention | Pre-intervention (day 1), post-intervention (day 4)
  A 26-item self-report questionnaire to measure social anxiety - Social Phobia and Anxiety Inventory for Children (SPAI-C; Biedel et al., 1998)

SECONDARY OUTCOMES:
Change from baseline in social anxiety at 2-week follow-up | Pre-intervention (day 1), 2-week follow-up post-intervention
  A 26-item self-report questionnaire to measure social anxiety - Social Phobia and Anxiety Inventory for Children (SPAI-C; Biedel et al., 1998)
Change from baseline in emotion sensitivity measurement at post-intervention and 2-week follow-up | Pre-intervention (day 1), post-intervention (day 4), 2-week follow-up post-intervention
  Emotion sensitivity measurement via shift in balance points across training sessions and at 2-week follow-up assessed using accuracy data from baseline and test phases of the ER/placebo training task
Change from baseline in fear of negative evaluation at post-intervention and 2-week follow-up | Pre-intervention (day 1), post-intervention (day 4), and 2-week follow-up
  A 12-item self-report questionnaire to measure fear of negative evaluation - Brief Fear of Negative Evaluation Questionnaire -Revised (BFNE-R; Carleton et al., 2006)
Change from baseline in anxiety related disorders at post-intervention and 2-week follow-up | Pre-intervention (day 1), post-intervention (week 4), and 2-week follow-up
  A 41-item self-report screening tool for anxiety disorders including panic, separation anxiety, generalized anxiety, social avoidance, and school phobia - Screen for Child Anxiety Related Disorders Child Version (SCARED; Birmaher et al., 1999)
Change from baseline in depression symptoms at post-intervention and 2-week follow-up | Pre-intervention (day 1), post-intervention (day 4), and 2-week follow-up
  A 10-item self-report subscale to assess the frequency of depressive symptoms - The Revised Child Anxiety and Depression Scale - Depression Subscale (RCADS; Chorpita et al., 2000)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Fitzgerald, PhD, Principal Investigator — University College Dublin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adams S, Penton-Voak IS, Harmer CJ, Holmes EA, Munafo MR. Effects of emotion recognition training on mood among individuals with high levels of depressive symptoms: study protocol for a randomised controlled trial. Trials. 2013 Jun 1;14:161. doi: 10.1186/1745-6215-14-161. PMID 23725208
- [Background] Penton-Voak IS, Bate H, Lewis G, Munafo MR. Effects of emotion perception training on mood in undergraduate students: randomised controlled trial. Br J Psychiatry. 2012 Jul;201(1):71-2. doi: 10.1192/bjp.bp.111.107086. Epub 2012 Apr 26. PMID 22539781
- [Background] Penton-Voak IS, Thomas J, Gage SH, McMurran M, McDonald S, Munafo MR. Increasing recognition of happiness in ambiguous facial expressions reduces anger and aggressive behavior. Psychol Sci. 2013 May;24(5):688-97. doi: 10.1177/0956797612459657. Epub 2013 Mar 26. PMID 23531485
- [Background] Yoon KL, Zinbarg RE. Threat is in the eye of the beholder: social anxiety and the interpretation of ambiguous facial expressions. Behav Res Ther. 2007 Apr;45(4):839-47. doi: 10.1016/j.brat.2006.05.004. Epub 2006 Jun 23. PMID 16797485
- [Background] Button K, Lewis G, Penton-Voak I, Munafo M. Social anxiety is associated with general but not specific biases in emotion recognition. Psychiatry Res. 2013 Nov 30;210(1):199-207. doi: 10.1016/j.psychres.2013.06.005. Epub 2013 Jul 9. PMID 23845415
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Wittchen HU, Fehm L. Epidemiology and natural course of social fears and social phobia. Acta Psychiatr Scand Suppl. 2003;(417):4-18. doi: 10.1034/j.1600-0447.108.s417.1.x. PMID 12950432
- [Background] Wittchen HU, Carter RM, Pfister H, Montgomery SA, Kessler RC. Disabilities and quality of life in pure and comorbid generalized anxiety disorder and major depression in a national survey. Int Clin Psychopharmacol. 2000 Nov;15(6):319-28. doi: 10.1097/00004850-200015060-00002. PMID 11110007
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition. Arlington, VA, American Psychiatric Association, 2013.
- [Background] Neil AL, Christensen H. Efficacy and effectiveness of school-based prevention and early intervention programs for anxiety. Clin Psychol Rev. 2009 Apr;29(3):208-15. doi: 10.1016/j.cpr.2009.01.002. Epub 2009 Jan 25. PMID 19232805
- [Background] Otto MW, Smits JA, Reese HE. Cognitive-behavioral therapy for the treatment of anxiety disorders. J Clin Psychiatry. 2004;65 Suppl 5:34-41. PMID 15078117
- [Background] Carleton RN, McCreary DR, Norton PJ, Asmundson GJ. Brief fear of negative evaluation scale-revised. Depress Anxiety. 2006;23(5):297-303. doi: 10.1002/da.20142. PMID 16688736
- [Background] Birmaher B, Brent DA, Chiappetta L, Bridge J, Monga S, Baugher M. Psychometric properties of the Screen for Child Anxiety Related Emotional Disorders (SCARED): a replication study. J Am Acad Child Adolesc Psychiatry. 1999 Oct;38(10):1230-6. doi: 10.1097/00004583-199910000-00011. PMID 10517055
- [Background] Crocetti E, Hale WW 3rd, Fermani A, Raaijmakers Q, Meeus W. Psychometric properties of the Screen for Child Anxiety Related Emotional Disorders (SCARED) in the general Italian adolescent population: a validation and a comparison between Italy and The Netherlands. J Anxiety Disord. 2009 Aug;23(6):824-9. doi: 10.1016/j.janxdis.2009.04.003. Epub 2009 Apr 23. PMID 19427168
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Mathyssek CM, Olino TM, Hartman CA, Ormel J, Verhulst FC, Van Oort FV. Does the Revised Child Anxiety and Depression Scale (RCADS) measure anxiety symptoms consistently across adolescence? The TRAILS study. Int J Methods Psychiatr Res. 2013 Mar;22(1):27-35. doi: 10.1002/mpr.1380. Epub 2013 Mar 11. PMID 23483654
- [Background] Beidel DC, Turner SM, Morris The Social Phobia and Anxiety Inventory for Children (SPAI-C). Toronto, ON, Multi-Health Systems, 1998.
- [Background] Inderbitzen-Nolan H, Davies CA, McKeon ND. Investigating the construct validity of the SPAI-C: comparing the sensitivity and specificity of the SPAI-C and the SAS-A. J Anxiety Disord. 2004;18(4):547-60. doi: 10.1016/S0887-6185(03)00042-2. PMID 15149713
- [Derived] Rawdon C, Murphy D, Motyer G, Munafo MR, Penton-Voak I, Fitzgerald A. An investigation of emotion recognition training to reduce symptoms of social anxiety in adolescence. Psychiatry Res. 2018 May;263:257-267. doi: 10.1016/j.psychres.2018.02.023. Epub 2018 Feb 8. PMID 29602534